CLINICAL TRIAL: NCT04921501
Title: Evaluation of Electrocardiographic Measurements by High Density Electrode ECG
Acronym: ECG-HD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2020/59
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Ventricular Arrhythmias
Keywords: Signal Averaging ECG; Cardiac electrophysiology

STUDY DESIGN:
Intervention Model Description: Prospective single arm monocentric descriptive and evaluation study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Proven or suspected arrhythmias group (Experimental)
  Interventions: Device: HD ECG; Device: Conventional 12-lead ECG

INTERVENTIONS:
Device: HD ECG — This experimental procedure is a passive, non-invasive, high-density surface ECG recording using 128 skin electrodes.The electrodes are positioned on strips of 10 electrodes to be prepared with adhesive tape and coated with conductive gel before installation on the patient. The total duration of the acquisition is 10 to 30 minutes.
Device: Conventional 12-lead ECG — This standard 12-lead ECG is defined on the HD ECG, from electrodes F13, G3, G14, H5, H15, H25 corresponding to the precordial electrodes. 4 limb electrodes will be added for the frontal leads. Thus, the HD and 12-lead ECGs will be obtained simultaneously.

SUMMARY:
Cardiac electrical activity is detected on the body surface with conventional electrocardiography involving 12 leads (ECG 12). A limitation of the current ECG technique is that recordings are obtained from only 6 independent precordial leads pairs ; which may miss cardiac potentials from spatially limited regions. More extensive sampling of the body surface may contribute to additional clinical information. The present study investigates the additional sensitivity of ECG using 128 body surface leads (High Density (HD) ECG) in measuring global or regional cardiac activity.

ELIGIBILITY:
Inclusion Criteria:

* Patient managed at the Bordeaux University Hospital for assessment of documented severe ventricular arrhythmia (VF, sudden resuscitated death) or suspected (syncope, family history of sudden death, ECG or Holter abnormality) or impaired ventricular conduction, OR
* Patients managed for prophylactic ventricular defibrillator implantation, according to international recommendations: Heart disease with ejection fraction < 35%, heart disease with sustained ventricular tachycardia, cardiomyopathies with high rhythmic risk,
* Women of childbearing age with effective contraception.

Exclusion Criteria:

* patients under 14 years old,
* pregnant or nursing woman.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2021-04-06 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Identification of the "amplitude" electrical criteria by HD ECG | Day 0
  These electrical criteria are measured in millivolt (mV)
Identification of the "cardiac time" electrical criteria by HD ECG | Day 0
  Defined by the auricular cardiac time, ventricular depolarization and repolarization time
Identification of the "duration" electrical criteria by HD ECG | Day 0
  These criteria are measured in milliseconds (ms)
Identification of "anatomical locations" electrical criteria by HD ECG | Day 0
  Defined by the position of the electrodes

CONTACTS AND LOCATIONS:
Overall Officials: Michel HAÏSSAGUERRE, MD-PhD, Principal Investigator — University Hospital, Bordeaux
Locations (11):
- France (10):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Privé Jacques Cartier, Massy
  - Hôpital Pitié-Salpêtrière, Paris
  - Hôpital Bichat, Paris
  - Hôpital européen Georges Pompidou, Paris
  - Bordeaux University Hospital, Pessac
  - CHR Pontchaillou, Rennes
  - CHU de Saint-Etienne, Saint-Etienne
  - CHU de Toulouse, Toulouse
  - CHU de Nancy, Vandœuvre-lès-Nancy
- Centre Hospitalier Princesse Grace, Monaco, Monaco